CLINICAL TRIAL: NCT04248738
Title: Social Needs and Resources in the Evaluation and Enhancement of Discharge Support: The NEEDS Study
Brief Title: Social Needs and Resources in the Evaluation and Enhancement of Discharge Support
Acronym: NEEDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Wallace (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Andrea Wallace, Associate Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00126445
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Social Determinants of Health; Readiness for Hospital Discharge
MeSH Terms: interventions — Health Services Needs and Demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SocNSuppR (Experimental): Inpatient teams systematically provided with information about patients' social needs and supportive resources.
  Interventions: Behavioral: NEEDS

INTERVENTIONS:
Behavioral: NEEDS — NEEDS intervention includes assessing patients' social needs and resources (SocNSuppR) and communicating those SocNSuppR to discharge teams

SUMMARY:
The goal of NEEDS is to systematically identify patients' needs and resources at home to inform discharge planning by health care teams. We believe the process of conducting such an assessment during hospitalization will integrate the patient's voice and improve patient outcomes by improving the team communication, quality of discharge planning, length of stay, post-discharge outcomes (e.g., satisfaction), and readmissions.

DETAILED DESCRIPTION:
As much as $17 billion could be saved annually by identifying patients at risk for hospital readmission, and better supporting them during their "transitions" home. However, current interventions aiming to decrease readmissions are limited by the fact that the most frequently used risk models relying on clinical and administrative data fail to identify a significant number of patients readmitted. A potential reason for the limited power of models seeking to identify those at risk for readmission is that they fail to incorporate patientcentered factors associated with health outcomes. Research continues to document how social needs (e.g. food and housing insecurity) and supportive resources (e.g. instrumental social support) play important roles in health outcomes. Yet, while admissions assessment of social needs and supportive resources is required for JCAHO and CMS, our previous research identified that 1) conducting an assessment of patients' supportive resources (i.e. instrumental social support) reveals information important to discharge planning (e.g., living alone, poor relationships with providers) otherwise unknown by inpatient teams; 2) lack of agreement between patients and nurses regarding readiness for hospital discharge (personal status, knowledge, coping ability, and expected support) is associated with patient coping difficulties and readmissions; and 3) even in systems with dedicated discharge planners (e.g., RN case managers, LCSWs), health team members involved in discharge planning and education are frequently unaware of patients' social needs and supportive resources. These findings suggest that facilitating communication between patients, family members, and inpatient health care providers regarding patients' social needs and supportive resources will improve patient outcomes (e.g., readiness for hospital discharge, readmissions). However, we do not yet understand whether or how patients' social needs and supportive resources inform clinical decision-making, and there are concerns about incorporating such assessments into routine care without sufficient understanding of its impact on patients. Therefore, the objective of this study is to provide inpatient health care teams with information about patients' social needs and supportive resources, evaluating whether it facilitates clinical decision-making, impacts readiness for hospital discharge and, ultimately, reduces hospital readmission. We will use a pre-post design, with a segmented regression (interrupted time series) analytic approach, to test the effect of communicating results of a SocNSuppR assessment to medical and surgical inpatient teams during routine discharge planning rounds, or the NEEDS intervention. The hypothesis is the incorporation of patients' SocNSuppR information into inpatient care will result in higher and more congruent readiness for hospital discharge ratings (between patients, family caregivers, and members of the health care team) compared to patients without SocNSuppR assessment and communication. The study's specific aims are:

Specific Aim 1. To test the effect of the NEEDS intervention (assessing patients' SocNSuppR and communicating SocNSuppR to discharge teams) on patient- family caregiver- nurse- provider- outcomes.

We will compare the following pre and post intervention: (1a) patient-reported readiness for hospital discharge (primary outcome) and post-discharge coping difficulty (secondary outcome), (1b) degree of congruence among readiness for hospital discharge ratings (among patients, families, caregivers, nurses, and providers), and (1c) 7- and 30-day readmission rates.

Specific Aim 2. To test the effect of the NEEDS intervention on discharge planning processes.

We will (2a) track changes in discharge plans based on SocNSuppR qualitatively through clinical documentation, and (2b) compare documentation of designated caregiver teaching, discharges before 11am, discharges before 2pm, time from discharge order to discharge, and HCAHPS scores.

Specific Aim 3. To examine patient and provider experiences of the NEEDS intervention.

We will qualitatively examine patient- caregiver- and provider-reported barriers, facilitators and recommendations for clinical adoption of the NEEDS protocol (SocNSuppR assessment and communication).

ELIGIBILITY:
Inclusion Criteria:

* newly assigned to one of the participating SS or GIM teams at the University Hospital

Exclusion Criteria:

* Non-English and non-Spanish speaking
* admitted due to a primary or secondary psychiatric diagnosis
* enrolled in palliative/hospice care
* unable to communicate verbally
* resident of skilled nursing facility upon admission
* transplant patient
* unfunded end stage renal disease patient
* incarcerated persons
* patients in isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4562 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Readiness for Hospital Discharge Scale (RHDS) | The RHDS is administered to all patients and clinical care team members for three months prior to the introduction of the intervention (baseline) and also during the 3-month intervention.
  Comparison of baseline and intervention average score on the Readiness for Hospital Discharge Scale, analyzed at the unit and hospital level. There are 8 questions on the RHDS, each scored from 0-10, with 0 indicating not being ready for discharge at all and 10 indicating being totally ready for discharge. Higher scores indicate better outcomes. The RHDS is administered to patients and the clinical care teams at the time that the patient receives the green light for discharge.

SECONDARY OUTCOMES:
Post-Discharge Coping Difficulty Scale (PDCDS) | The PDCDS is administered to all patients for three months prior to the introduction of the intervention (baseline) and also during the 3-month intervention.
  Comparison of baseline and intervention average score on the Post-Discharge Coping Difficulty Scale, analyzed at the unit and hospital level. There are 10 questions on the RHDS, each scored from 0-10, with 0 indicating no difficulty coping with life after discharge and 10 indicating a great deal of difficulty coping. Higher scores indicate worse outcomes. The RHDS is only administered to patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallace AS, Park S, Guo JW, Johnson EP, Elliott M, Elmore CE, Bristol AA. Reconsidering risk: instrumental social support and 30-day utilization after discharge. Health Aff Sch. 2025 Sep 4;3(10):qxaf178. doi: 10.1093/haschl/qxaf178. eCollection 2025 Oct. PMID 41079423
- [Derived] Wallace AS, Raaum SE, Johnson EP, Presson AP, Allen CM, Elliott M, Bristol AA, Elmore CE. Impact of COVID-19 visitation policies and hospital capacity on discharge readiness in medicine patients. Discov Health Syst. 2023;2(1):45. doi: 10.1007/s44250-023-00060-8. Epub 2023 Nov 30. PMID 38045443
- [Derived] Schmutz KE, Wallace AS, Bristol AA, Johnson EP, Raaum SE. Hospital Discharge During COVID-19: The Role of Social Resources. Clin Nurs Res. 2022 May;31(4):724-732. doi: 10.1177/10547738221075760. Epub 2022 Feb 15. PMID 35168380